CLINICAL TRIAL: NCT06750471
Title: Efficacy of Alternate Dupilumab Schedule in Recurrent Chronic Rhinosinusitis With Nasal Polyposis Patients
Brief Title: Dupixent Study for Alternate Administration
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Collaborators: Tripler Army Medical Center (U.S. Federal Agency); Fort Belvoir Community Hospital (U.S. Federal Agency); William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222008
Record Dates: First submitted 2021-08-30; First posted 2024-12-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Nasal Polyps; Sinusitis; Chronic Disease
Keywords: Chronic rhinosinusitis; Dupilumab; Biologic Therapy
MeSH Terms: conditions — Nasal Polyps; Sinusitis; Chronic Disease | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Regular Adminstration (Active Comparator): Eligible patient will receive 300 mg Subcutaneous Dupilumab every 2 weeks for 28 weeks
  Interventions: Biological: Dupilumab
- Arm B - Alternate Administration (Experimental): Eligible patient will receive 300 mg Subcutaneous Dupilumab every 2 weeks for 8 weeks and then every 4 weeks up until 28 weeks
  Interventions: Biological: Dupilumab

INTERVENTIONS:
Biological: Dupilumab — Dupilumab is an anti-IL 4-13 biologic therapy that has been recently approved for use in recurrent chronic rhinosinusitis with nasal polyposis.
  Other Names: Dupixent

SUMMARY:
Investigators will investigate an alternate Dupilumab administration schedule in patients with recurrent chronic rhinosinusitis with nasal polyposis, who have a history of full endoscopic sinus surgery and are on appropriate topical medical therapies. Specifically, investigators will investigate if the alternate schedule of drug administration is non-inferior in both subjective and objective outcomes.

DETAILED DESCRIPTION:
Dupixent was recently approved by the FDA for chronic rhinosinusitis patients with nasal polyposis in April 2019. Literature support for this approval comes from results obtained from a landmark Phase III trial (LIBERTY SINUS-24 and SINUS-52) that were published in November 2019. The data suggests that Dupilumab improves subjective quality of life significantly in patients with chronic sinusitis with nasal polyposis and there is objective evidence of decreased disease burden and severity of other comorbidities (asthma, aspirin exacerbated respiratory disease). Therefore, there is robust scientific evidence supporting the use of this medication in chronic rhinosinusitis with nasal polyposis patients along with the FDA indication for usage of this medication in this subset of patients.

Otolaryngologists see and manage most (if not all) of chronic sinusitis patients with persistent symptoms and give recommendations for surgical and medical therapies. Given our unique ability to perform a detailed examination and provide medical and surgical care, investigators believe that this patient population will be best served with us making the determination of when to initiate the treatment if other treatment strategies fail. Given the cost associated with this medication (~ $45,630/patient/year based on price of $1,755/injection), investigators can make the judicious determination for when to prescribe this medication based on published evidence and guidelines in literature.

After careful assessment of LIBERTY study, most subjective and objective outcomes appear to show statistically and clinically significant benefit after 8 weeks of therapy. Moreover, one of the study arms had patients on this medication every 2 weeks until 26 weeks and then switched to every 4 weeks for the rest of the year. Given the apparent benefit of medication compared to placebo at 8 weeks, investigators propose that an alternate medication schedule with less frequent dosing after 8 weeks will be just as effective in improving subjective and objective outcomes in this patient population. If a non-inferior improvement is noted in the alternate medication schedule, then this will translate into significant cost saving to DoD and DHA (~$21,000/patient/year) when patients are placed on this medication due to the refractory nature of their disease.

Moreover, if the alternate schedule is just as effective, then this will validate use of this schedule in active duty service members (ADSM) during temporary duty or deployments to keep them medically fit and ready. Although topical steroid rinses are beneficial after surgery, the lack of distilled water in some austere environments prohibit usage and some patients have disease recurrence despite steroids and therefore require alternate medications or additional surgery. If the alternate regimen is proven to be non-inferior, then ADSMs or their medical team can carry the pre-made medication with them while following appropriate storage instructions according to drug information. Based on the FDA information website, Dupilumab can be stored below the room temperature (<77F or <25C) in pre-filled syringes up to 14 days or within refrigerator (between 2-8 C) until expiration. As long as these storage conditions can be met, ADSMs can continue this regimen while they are away. Additionally, if they are stable on long term Dupilumab therapy, there is potential for even longer time intervals between injections to help manage their chronic disease process.

ELIGIBILITY:
Eligibility: patients =>18 years old with recurrent chronic rhinosinusitis with nasal polyposis (CRSwNP) despite standard of care (i.e topical medical therapies and full endoscopic sinus surgery)

Inclusion criteria:

* Age=>18 y/o with recurrent CRSwNP based on reported symptoms and endoscopic assessment
* history of atleast 1 endoscopic sinus surgery
* Current use of intranasal corticosteroid spray or irrigation
* Active duty servicemembers must be in the area for at least 7 months after starting the medication to complete the necessary follow ups

Exclusion Criteria:

* Previous use of other biologic therapy in last 6 months
* if history of asthma, FEV1< 50%
* history of cystic fibrosis, eosinophilic granulomatosis with polyangiitis, granulomatosis with polyangiitis, kartagener syndrome, primary ciliary dyskinesia
* Patient is a pregnant woman, may become pregnant or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Sinonasal outcome test - 22 over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  22 item questionnaire of impact of chronic rhinosinusitis on quality of life. Scored from 0-120: higher number = worse symptoms
Change in Lund Kennedy Score over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  Sinus endoscopy to objectively score the impact of drug on patient's disease process. Total points = 20 (10 on each side), higher score = worse objective data
Change in Total polyp score over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  Sinus endoscopy to objectively score the impact of drug on patient's disease process. Scored from 0-8, 4 on each side. Higher scores = worse polyp scores
Change in Rhinosinusitis Disability Index Score (RSDI) over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  Disability associated with chronic rhinosinusitis, Scored from 0-120: higher number = worse quality of life.

SECONDARY OUTCOMES:
Change in IgE levels over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  Labs to evaluate the impact of Dupilimab administration in patients
Change in Eosinophil levels over different time intervals | Baseline, week 4, week 8, week 16 and week 28
  Labs to evaluate the impact of Dupilimab administration in patients
Cost Savings between 2 treatment arms | Ove the course of the study timeline - 28 weeks
  Cost savings between the two treatment arms will be compared to see how cost to healthcare was saved with alternate therapy.
Need for additional interventions or surgeries in each arm | Over the course of the study timeline - 28 weeks
  We will assess if participants needed oral steroids or surgeries while being on dupixent therapy over the course of study to help manage their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Renee M Serra, MD, Principal Investigator — ENT/Audiology Department Chair; Roy F Thomas, MD, Principal Investigator — Rhinologist
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The IPD information will only be available to the researchers participating in this multi-site trial. No outside researcher will be able to view this data or information.

REFERENCES:
- [Background] Bachert C, Han JK, Desrosiers M, Hellings PW, Amin N, Lee SE, Mullol J, Greos LS, Bosso JV, Laidlaw TM, Cervin AU, Maspero JF, Hopkins C, Olze H, Canonica GW, Paggiaro P, Cho SH, Fokkens WJ, Fujieda S, Zhang M, Lu X, Fan C, Draikiwicz S, Kamat SA, Khan A, Pirozzi G, Patel N, Graham NMH, Ruddy M, Staudinger H, Weinreich D, Stahl N, Yancopoulos GD, Mannent LP. Efficacy and safety of dupilumab in patients with severe chronic rhinosinusitis with nasal polyps (LIBERTY NP SINUS-24 and LIBERTY NP SINUS-52): results from two multicentre, randomised, double-blind, placebo-controlled, parallel-group phase 3 trials. Lancet. 2019 Nov 2;394(10209):1638-1650. doi: 10.1016/S0140-6736(19)31881-1. Epub 2019 Sep 19. PMID 31543428
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Fokkens WJ, Lund V, Bachert C, Mullol J, Bjermer L, Bousquet J, Canonica GW, Deneyer L, Desrosiers M, Diamant Z, Han J, Heffler E, Hopkins C, Jankowski R, Joos G, Knill A, Lee J, Lee SE, Marien G, Pugin B, Senior B, Seys SF, Hellings PW. EUFOREA consensus on biologics for CRSwNP with or without asthma. Allergy. 2019 Dec;74(12):2312-2319. doi: 10.1111/all.13875. Epub 2019 Jul 15. PMID 31090937
- [Background] Bachert C, Mannent L, Naclerio RM, Mullol J, Ferguson BJ, Gevaert P, Hellings P, Jiao L, Wang L, Evans RR, Pirozzi G, Graham NM, Swanson B, Hamilton JD, Radin A, Gandhi NA, Stahl N, Yancopoulos GD, Sutherland ER. Effect of Subcutaneous Dupilumab on Nasal Polyp Burden in Patients With Chronic Sinusitis and Nasal Polyposis: A Randomized Clinical Trial. JAMA. 2016 Feb 2;315(5):469-79. doi: 10.1001/jama.2015.19330. PMID 26836729
- [Background] Van Crombruggen K, Zhang N, Gevaert P, Tomassen P, Bachert C. Pathogenesis of chronic rhinosinusitis: inflammation. J Allergy Clin Immunol. 2011 Oct;128(4):728-32. doi: 10.1016/j.jaci.2011.07.049. Epub 2011 Aug 24. PMID 21868076
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Senior BA, Glaze C, Benninger MS. Use of the Rhinosinusitis Disability Index (RSDI) in rhinologic disease. Am J Rhinol. 2001 Jan-Feb;15(1):15-20. doi: 10.2500/105065801781329428. PMID 11258649